CLINICAL TRIAL: NCT01978236
Title: An Open-Label, Multicentre, Corollary Study of Pre-Operative Therapy With Dabrafenib and the Combination of Dabrafenib With Trametinib in Subjects With BRAF Mutation-Positive Metastatic Melanoma to the Brain
Brief Title: Dabrafenib/Trametinib, BRAF or BRAF AND MEK Pre-op With BRAF and MEK Post-op, Phase IIB, Melanoma With Brain Mets,Biomarkers and Metabolites
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to the limited enrollment.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116521
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Melanoma and Brain Metastases
Keywords: BRAF V600E mutation; brain metastases; BRAF V600K mutation; Metastatic melanoma; BRAF inhibitor; brain neoplasms; GSK2118436
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): The first cohort of 15 subjects will receive oral dabrafenib 150 mg twice daily orally for 7 to 14 days prior to surgery in Cohort A; Subjects will be treated for at least 7 days prior to craniotomy, but not more than 14 days. Subjects in either cohort with intracranial and/or extracranial metastases remaining after surgery may resume treatment with the combination of dabrafenib 150 mg BID and trametinib 2 mg once daily no earlier than 72 hours after surgery
  Interventions: Drug: Dabrafenib 150 mg
- Cohort B (Experimental): The second cohort of 15 subjects will receive dabrafenib 150 mg twice daily combined with trametinib 2 mg once daily (Cohort B) orally for 7 to 14 days prior to surgery; Subjects will be treated for at least 7 days prior to craniotomy, but not more than 14 days. Subjects in either cohort with intracranial and/or extracranial metastases remaining after surgery may resume treatment with the combination of dabrafenib 150 mg BID and trametinib 2 mg once daily no earlier than 72 hours after surgery
  Interventions: Drug: Dabrafenib 150 mg; Drug: Trametinib 2.0 mg

INTERVENTIONS:
Drug: Dabrafenib 150 mg — Dabrafenib will be provided for oral administration as 50 mg and 75 mg capsules. Dabrafenib will be dosed orally with approximately 200 mL of water, twice a day. Dabrafenib should be administered under fasting conditions.
Drug: Trametinib 2.0 mg — Trametinib study treatment will be provided as 0.5 mg and 2.0 mg tablets. should be taken orally with approximately 200 mL of water under fasting conditions, either one hour before or two hours after a meal.
  Arms: Cohort B

SUMMARY:
This is a global, multi-centre, open-label, study of GSK2118436 conducted in up to 30 evaluable subjects with resectable, BRAF V600E or V600K mutation-positive metastatic melanoma to the brain. All subjects in this study are required to have accessible extracranial metastases and are agreeable to undergo repetitive biopsies. The first cohort of 15 subjects will receive dabrafenib orally 150mg twice daily (BID) for 7 to 14 days prior to surgery (Cohort A); the second cohort of 15 subjects will receive the combination of dabrafenib 150 mg BID and trametinib 2 mg once daily for 7 to 14 days prior to surgery (Cohort B). The primary purpose of this study is to determine levels and distribution of dabrafenib, its metabolites, and trametinib (Cohort B only) in parenchymal brain metastases, extracranial metastases, and peripheral blood (plasma) within two cohorts of subjects with BRAF V600E/K mutation-positive melanoma that has metastasized to the brain. All subjects will be followed for survival and new anti-cancer therapy for a total of two years or until death or the subject wishes to withdraw from further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically-confirmed metastatic melanoma (Stage IV), carrying BRAF V600E or V600K mutation as determined by testing certified for clinical diagnostic purposes. Previously performed certified BRAF testing is acceptable. If no prior BRAF mutation testing results are available, testing of a distant metastasis is preferred, but testing of a regional metastasis or primary tumor is also acceptable
* At least one intracranial lesion >=1.0 cm but <=4.0 cm that can be treated with surgical resection in the opinion of the treating physicians, and for which immediate local therapy is not clinically indicated
* At least two extracranial lesions that are easily accessible for biopsy, in the judgment of the treating physician. Easily accessible tumors may include cutaneous, subcutaneous, and superficial lymph node metastases.
* Age >18 years of age.
* Able to swallow and retain oral medication
* Women with child-bearing potential must be willing to practice acceptable methods of birth control during the study
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment.
* Must be able to understand and comply with protocol requirements and instructions
* Eastern Co-operative Oncology Group (ECOG) performance status of 0-2
* Must have adequate organ function as defined by the following screening values (Retesting of borderline screening organ function and treatment with blood transfusions, growth factors etc. will be allowed):
* Absolute neutrophil count (ANC) >=1.2x10^9/L
* Hemoglobin >=9 g/dL
* Platelets >=100x10^9/L
* Serum bilirubin <=1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5xULN
* Serum creatinine <=1.5 mg/dL (If serum creatinine is >1.5 mg/dL, calculate creatinine clearance using standard Cockcroft and Gault Method Creatinine clearance must be >50 mL/min)
* Prothrombin time (PT)/International normalized ratio (INR) and partial thromboplastin time (PTT) <=1.3xULN
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN)

Exclusion Criteria:

* Neurological symptoms related to brain metastasis that are not controlled with a stable or decreasing dose of oral steroids for at least 7 days prior to starting GSK2118436
* Prior Central Nervous System (CNS)-directed local therapies, including surgical resection, whole brain radiation (WBRT), Stereotactic radiosurgery (SRS), or gamma knife (GK)
* Previous treatment with a BRAF or MEK inhibitor
* Cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) or investigational anti-cancer drugs within the last 3 weeks, or chemotherapy without delayed toxicity within the last 2 weeks, preceding the first dose of study treatment.
* Current or expected use of a prohibited medication, including enzyme-inducing antiepileptic drugs (EIAEDs) during treatment with GSK2118436.
* Presence of leptomeningeal disease or dural metastases.
* History of another active malignancy within the past 5 years, or any malignancy with a confirmed activating RAS mutation. The prospective RAS mutation testing is not required, however, if results of previous RAS testing are known, they must be used in assessing eligibility. Subjects with a history of completely resected non-melanoma skin cancer are eligible.
* Known allergies against contrast agents required for magnetic resonance imaging (MRI) of intracranial lesions, or other contraindications for MRI, i.e., pacemaker
* Current use of therapeutic warfarin. Low-molecular-weight heparin and prophylactic low-dose warfarin are permitted
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0) Grade 2 or higher from previous anti-cancer therapy, except alopecia
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs.
* History of a prior symptomatic stroke, dementia, or other significant central neurologic condition (i.e. multiple sclerosis)
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
* Current acute infection requiring intravenous antibiotics
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* The history or evidence of following cardiac abnormalities:
* Corrected QT (QTc) interval using Bazett's Formula; (QTcB) >= 480 msecs
* A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
* Coronary angioplasty or stenting within the past 12 weeks
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Abnormal cardiac valve morphology (>= Grade 2) documented by echocardiogram (ECHO)
* History of or evidence of clinically significant uncontrolled cardiac arrhythmias
* Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic >90 mm Hg which cannot be controlled by anti-hypertensive therapy
* Subjects with intra-cardiac defibrillators or permanent pacemakers
* Pregnant, lactating or breastfeeding females
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2118436 or excipients that contraindicate their participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (2):
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, North Sydney, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six participants (five male and one female) with resectable, BRAF V600E or V600K mutation-positive metastatic melanoma to the brain were enrolled into the study, all into Cohort A. There were no participants enrolled in Cohort B.
Groups:
- Cohort A: Participants in Cohort A received dabrafenib orally 150 milligram twice daily for 7 to 14 days prior to surgery.
Period: Overall Study
Arm/Group | Cohort A
Started | 6
Completed | 4
Not Completed | 2
Not completed — Discontinued due to study close | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (16.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African Heritage | 1
  White/Caucasian/European Heritage | 5

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Dabrafenib, Its Metabolites Hydroxy-, Carboxy- and Desmethyl-dabrafenib in Peripheral Blood (Plasma)
Description: Blood samples for pharmacokinetic analysis of dabrafenib and its active metabolites, including hydroxy-, carboxy-, and desmethyl-dabrafenib were collected on day of surgical resection of the brain metastasis(es), Two samples were collected before surgery and 2 samples after surgery with one hour gap in between. Upon collection blood was placed on wet ice. Plasma was isolated within 60 minutes of collection and frozen at -20 degree celsius.
Time Frame: Pre-surgery and post-surgery on Day 15
Population: The Pharmacokinetic analysis set included all participants who provided at least one evaluable Pharmacokinetic concentration.
Measure: Number; unit: Nano grams per milliliter (ng/mL)
Arm/Group | Cohort A
Number analyzed (Participants) | 6
Nano grams per milliliter (ng/mL)
  Participant 1, Dabrafenib, Pre-Surgery 1 | 2.54
  Participant 1, Dabrafenib, Pre-Surgery 2 | 2.66
  Participant 1, Dabrafenib, Post-Surgery 1 | 1.24
  Participant 1, Dabrafenib, Post-Surgery 2 | 1.32
  Participant 1, Desmethyl-dabrafenib,Pre-Surgery 1 | 357
  Participant 1, Desmethyl-dabrafenib,Pre-Surgery 2 | 438
  Participant 1, Desmethyl-dabrafenib,Post-Surgery 1 | 153
  Participant 1, Desmethyl-dabrafenib,Post-Surgery 2 | 147
  Participant 1,Hydroxy-dabrafenib,Pre-Surgery 1 | 4.72
  Participant 1,Hydroxy-dabrafenib,Pre-Surgery 2 | 4.91
  Participant 1,Hydroxy-dabrafenib,Post-Surgery 1 | 1.66
  Participant 1,Hydroxy-dabrafenib,Post-Surgery 2 | 1.58
  Participant 1,carboxy-dabrafenib,Pre-Surgery 1 | 694
  Participant 1,carboxy-dabrafenib,Pre-Surgery 2 | 621
  Participant 1,carboxy-dabrafenib,Post-Surgery 1 | 454
  Participant 1,carboxy-dabrafenib,Post-Surgery 2 | 423
  Participant 2, Dabrafenib, Pre-Surgery 1 | 953
  Participant 2, Dabrafenib, Pre-Surgery 2 | 596
  Participant 2, Dabrafenib, Post-Surgery 1 | 137
  Participant 2, Dabrafenib, Post-Surgery 2 | 119
  Participant 2, Desmethyl-dabrafenib,Pre-Surgery 1 | 150
  Participant 2, Desmethyl-dabrafenib,Pre-Surgery 2 | 180
  Participant 2, Desmethyl-dabrafenib,Post-Surgery 1 | 90.1
  Participant 2, Desmethyl-dabrafenib,Post-Surgery 2 | 79.1
  Participant 2,Hydroxy-dabrafenib,Pre-Surgery 1 | 644
  Participant 2,Hydroxy-dabrafenib,Pre-Surgery 2 | 507
  Participant 2,Hydroxy-dabrafenib,Post-Surgery 1 | 102
  Participant 2,Hydroxy-dabrafenib,Post-Surgery 2 | 101
  Participant 2,carboxy-dabrafenib,Pre-Surgery 1 | 2010
  Participant 2,carboxy-dabrafenib,Pre-Surgery 2 | 3020
  Participant 2,carboxy-dabrafenib,Post-Surgery 1 | 2150
  Participant 2,carboxy-dabrafenib,Post-Surgery 2 | 2040
  Participant 3, Dabrafenib, Pre-Surgery 1 | 151
  Participant 3, Dabrafenib, Pre-Surgery 2 | 127
  Participant 3, Dabrafenib, Post-Surgery 1 | 18.2
  Participant 3, Dabrafenib, Post-Surgery 2 | 12.6
  Participant 3, Desmethyl-dabrafenib,Pre-Surgery 1 | 532
  Participant 3, Desmethyl-dabrafenib,Pre-Surgery 2 | 656
  Participant 3, Desmethyl-dabrafenib,Post-Surgery 1 | 295
  Participant 3, Desmethyl-dabrafenib,Post-Surgery 2 | 238
  Participant 3,Hydroxy-dabrafenib,Pre-Surgery 1 | 215
  Participant 3,Hydroxy-dabrafenib,Pre-Surgery 2 | 182
  Participant 3,Hydroxy-dabrafenib,Post-Surgery 1 | 36.2
  Participant 3,Hydroxy-dabrafenib,Post-Surgery 2 | 24.9
  Participant 3,carboxy-dabrafenib,Pre-Surgery 1 | 4360
  Participant 3,carboxy-dabrafenib,Pre-Surgery 2 | 4300
  Participant 3,carboxy-dabrafenib,Post-Surgery 1 | 2620
  Participant 3,carboxy-dabrafenib,Post-Surgery 2 | 2570
  Participant 4, Dabrafenib, Pre-Surgery 1 | 134
  Participant 4, Dabrafenib, Pre-Surgery 2 | 111
  Participant 4, Dabrafenib, Post-Surgery 1 | 10.2
  Participant 4, Dabrafenib, Post-Surgery 2 | 6.84
  Participant 4, Desmethyl-dabrafenib,Pre-Surgery 1 | 896
  Participant 4, Desmethyl-dabrafenib,Pre-Surgery 2 | 961
  Participant 4, Desmethyl-dabrafenib,Post-Surgery 1 | 377
  Participant 4, Desmethyl-dabrafenib,Post-Surgery 2 | 286
  Participant 4,Hydroxy-dabrafenib,Pre-Surgery 1 | 106
  Participant 4,Hydroxy-dabrafenib,Pre-Surgery 2 | 86.1
  Participant 4,Hydroxy-dabrafenib,Post-Surgery 1 | 13.7
  Participant 4,Hydroxy-dabrafenib,Post-Surgery 2 | 9.54
  Participant 4,carboxy-dabrafenib,Pre-Surgery 1 | 1390
  Participant 4,carboxy-dabrafenib,Pre-Surgery 2 | 1380
  Participant 4,carboxy-dabrafenib,Post-Surgery 1 | 865
  Participant 4,carboxy-dabrafenib,Post-Surgery 2 | 620
  Participant 5, Dabrafenib, Pre-Surgery 1 | 101
  Participant 5, Dabrafenib, Pre-Surgery 2 | 51.1
  Participant 5, Dabrafenib, Post-Surgery 1 | 15.4
  Participant 5, Dabrafenib, Post-Surgery 2 | 11
  Participant 5, Desmethyl-dabrafenib,Pre-Surgery 1 | 661
  Participant 5, Desmethyl-dabrafenib,Pre-Surgery 2 | 420
  Participant 5, Desmethyl-dabrafenib,Post-Surgery 1 | 433
  Participant 5, Desmethyl-dabrafenib,Post-Surgery 2 | 386
  Participant 5,Hydroxy-dabrafenib,Pre-Surgery 1 | 312
  Participant 5,Hydroxy-dabrafenib,Pre-Surgery 2 | 183
  Participant 5,Hydroxy-dabrafenib,Post-Surgery 1 | 62.5
  Participant 5,Hydroxy-dabrafenib,Post-Surgery 2 | 52.4
  Participant 5,carboxy-dabrafenib,Pre-Surgery 1 | 4580
  Participant 5,carboxy-dabrafenib,Pre-Surgery 2 | 3750
  Participant 5,carboxy-dabrafenib,Post-Surgery 1 | 2770
  Participant 5,carboxy-dabrafenib,Post-Surgery 2 | 2550
  Participant 6, Dabrafenib, Pre-Surgery 1 | 176
  Participant 6, Dabrafenib, Pre-Surgery 2 | 106
  Participant 6, Dabrafenib, Post-Surgery 1 | 83.2
  Participant 6, Dabrafenib, Post-Surgery 2 | 61.4
  Participant 6, Desmethyl-dabrafenib,Pre-Surgery 1 | 1530
  Participant 6, Desmethyl-dabrafenib,Pre-Surgery 2 | 1050
  Participant 6, Desmethyl-dabrafenib,Post-Surgery 1 | 1310
  Participant 6, Desmethyl-dabrafenib,Post-Surgery 2 | 1200
  Participant 6,Hydroxy-dabrafenib,Pre-Surgery 1 | 326
  Participant 6,Hydroxy-dabrafenib,Pre-Surgery 2 | 227
  Participant 6,Hydroxy-dabrafenib,Post-Surgery 1 | 197
  Participant 6,Hydroxy-dabrafenib,Post-Surgery 2 | 151
  Participant 6,carboxy-dabrafenib,Pre-Surgery 1 | 2680
  Participant 6,carboxy-dabrafenib,Pre-Surgery 2 | 2250
  Participant 6,carboxy-dabrafenib,Post-Surgery 1 | 2170
  Participant 6,carboxy-dabrafenib,Post-Surgery 2 | 2410

2. Primary Outcome: Concentrations of Dabrafenib, Its Metabolites Hydroxy-, Carboxy- and Desmethyl-dabrafenib in Parenchymal Brain Metastases
Description: Concentrations of dabrafenib, its metabolites, hydroxy-, carboxy, and desmethyl-dabrafenib, and possibly other drug-related species were quantified in the pharmacokinetic tissue sample by an investigative Liquid chromatography- mass spectrometry (LC-MS)/MS method. The spatial distribution of dabrafenib, its metabolites, hydroxy-, carboxy, and desmethyl-dabrafenib and possibly other drug-related species in the tissue samples were determined using an investigative matrix assisted laser desorption ionization (MALDI) analysis method. Parenchymal brain metastases and extracranial metastases using MALDI imaging was not determined for all participants (completed by GSK for the first two participants enrolled)
Time Frame: Day 15
Population: Pharmacokinetic Analysis Set
Measure: Number; unit: ng/mL
Arm/Group | Cohort A
Number analyzed (Participants) | 6
ng/mL
  Participant 1,Dabrafenib | 0
  : Participant 1, Hydroxy-dabrafenib | 0
  Participant 1, Carboxy-dabrafenib | 131
  Participant 1, Desmethyl-dabrafenib | 60
  Participant 2,Dabrafenib | 57.0
  Participant 2, Hydroxy-dabrafenib | 16.0
  Participant 2, Carboxy-dabrafenib | 81.0
  Participant 2, Desmethyl-dabrafenib | 15.0
  Participant 3,Dabrafenib | 40.5
  Participant 3, Hydroxy-dabrafenib | 63.7
  Participant 3, Carboxy-dabrafenib | 628
  Participant 3, Desmethyl-dabrafenib | 53.4
  Participant 4,Dabrafenib | 0
  Participant 4, Hydroxy-dabrafenib | 0
  Participant 4, Carboxy-dabrafenib | 228
  Participant 4, Desmethyl-dabrafenib | 88.4
  Participant 5,Dabrafenib | 22.5
  Participant 5, Hydroxy-dabrafenib | 94.3
  Participant 5, Carboxy-dabrafenib | 898
  Participant 5, Desmethyl-dabrafenib | 82.3
  Participant 6,Dabrafenib | 124
  Participant 6, Hydroxy-dabrafenib | 261
  Participant 6, Carboxy-dabrafenib | 660
  Participant 6, Desmethyl-dabrafenib | 197

3. Primary Outcome: Concentrations of Dabrafenib, Its Metabolites Hydroxy-, Carboxy- and Desmethyl-dabrafenib) and Trametinib (Cohort B Only) in CSF Samples.
Description: Blood samples for pharmacokinetic analysis of dabrafenib and its active metabolites, including hydroxy-, carboxy-, and desmethyl-dabrafenib and trametinib (as appropriate), were planned but not collected.
Time Frame: Pre-surgery and post-surgery on Day 15
Population: Pharmacokinetic Analysis Set
Arm/Group | Cohort A
Number analyzed (Participants) | 0

4. Secondary Outcome: Concentrations of Dabrafenib, Its Metabolites Hydroxy-, Carboxy- and Desmethyl-dabrafenib) in Cerebrospinal Fluid (CSF) Samples
Description: Concentrations of dabrafenib, its metabolites hydroxy-, carboxy- and desmethyl-dabrafenib) and trametinib in CSF (in participants who agree for optional collection of CSF at the time of brain tumor resection). Optional collection of CSF was obtained in the operating room on the day of brain metastasis resection. CSF samples for only one participant were collected and analyzed.
Time Frame: Day 15
Population: Pharmacokinetic Analysis Set
Measure: Number; unit: ng/mL
Arm/Group | Cohort A
Number analyzed (Participants) | 1
ng/mL
  Dabrafenib | 0.00
  Desmethyl-dabrafenib | 2.30
  Hydroxy-dabrafenib | 2.26
  Carboxy-dabrafenib | 36.9

5. Secondary Outcome: Number of Participants With Changes in Mitogen-activated Protein Kinase (MAPK) Pathway Markers
Description: Changes in MAPK pathway markers in paired extracranial biopsies taken pre-treatment, during craniotomy, and at disease progression, and changes in markers between post-operative intracranial and extracranial biopsies was planned but not performed as the study was terminated due to low enrollment.
Time Frame: Up to Day 15
Population: Full Analysis Set. Analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Changes in Radiographic Tumors
Description: Changes in the radiographic characteristics of the tumors were planned to be compared to (1) levels of dabrafenib, its metabolites and trametinib (where appropriate) in the brain metastases, plasma, and CSF, and (2) MAPK pathway activation status in tumors at the time of surgery. Results were planned to be compared to the analysis of early clinical responses in extracranial metastases, as determined by the Positron emission tomography (PET-CT) imaging. This analysis was planned but not performed as the study was terminated due to low enrollment
Time Frame: Up to 2 years
Population: Full Analysis Set. Analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

7. Secondary Outcome: Percent Change From Baseline to Pre-surgery in the Sum of the Longest Diameters (SLD) of Intracranial Target Lesions
Description: The change from Baseline to the pre-surgery intracranial disease assessment in the SLD of intracranial target lesions was planned to be calculated as a percentage change from the baseline SLD. It was planned to be reported for the V600E and V600K analysis populations for each cohort and also aggregately if appropriate. This analysis was planned but not performed as the study was terminated due to low enrollment.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

8. Secondary Outcome: Maximum Percent Change From Baseline in the SLD of Unresected Intracranial Target Lesions
Description: The maximum change from Baseline in the SLD of unresected intracranial target lesions was planned to be calculated as a percentage change from the baseline SLD. It was planned to be reported for the V600E and V600K analysis populations for each cohort and also aggregately if appropriate. This analysis was planned but not performed as the study was terminated due to low enrollment.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants With Overall Extracranial Response Rate in Unresected Lesions
Description: Overall Extracranial Response Rate was defined as the percentage of participants with Complete response (CR) or Partial response (PR) at anytime as per modified Response Evaluation Criteria in Solid Tumors (RECIST). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence and is determined programmatically based on the investigator's assessment of response at each time point. Overall Extracranial Response Rate was planned but not analyzed as the study was terminated due to low enrollment.
Time Frame: Approximately 2 years or death whichever occurs first
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival, defined as the time from first dose of study treatment to death for any reason, was planned to summarize using Kaplan-Meier quartile estimates along with two sided 95% confidence intervals. But were not performed as the study was terminated due to low enrollment.
Time Frame: Approximately 2 years or death whichever occurs first
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital sign measurements including temperature, respiratory rate, systolic and diastolic blood pressure, and pulse rate were planned to be performed but were neither summarized nor listed as the study was terminated.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Abnormal Physical Examinations
Description: A complete physical examination was planned which included assessments of the head, eyes, ears, nose, throat, skin, thyroid, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes, and extremities. Height and weight was also planned to be measured and recorded. A complete physical exam including a thorough genitourinary examination for female participants, inspection of the head and neck region, and digital rectal examination for both male and female participants was planned to be performed at Screening, and Month 12 or at discontinuation if discontinuation occurs prior to Month 12. If the participants had a genitourinary and rectal exam within 6 months of screening, these assessments need not to be repeated at screening. But data for physical examinations were not summarized and listed as the study was terminated.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiograms (ECG)
Description: 112-lead ECGs were planned to be obtained at screening during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. At each assessment a 12-lead ECG was planned to be performed by qualified personnel at the site after at least a five-minute rest with the participants in a semi-recumbent or supine position. But data for 12-lead ECGs were not summarized and listed as the study was terminated.
Time Frame: Screening
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Abnormal Echocardiogram (ECHO)
Description: ECHO include an evaluation for Left ventricular ejection fraction (LVEF) and both right- and left-sided valvular lesions. ECHO was planned to be performed at screening, Week 8 and every 16 weeks till discontinuation. data for ECHO was not summarized and listed as the study was terminated.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Assessments
Description: Laboratory assessments included parameters like Hematology, Standard Chemistry, Coagulation, Serum Pregnancy. Assessment of these parameters were planned to be performed by the central laboratory on screening, Day prior to surgery, Every 4 weeks after restart and Discontinuation, but were not analyzed as the study was terminated due to low enrollment.
Time Frame: Up to 2 years
Population: Full Analysis Set. This analysis was planned but not performed as the study was terminated due to low enrollment.
Arm/Group | Cohort A
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE were collected from the time the first dose of study treatment is administered until 30 days following discontinuation of study treatment regardless of initiation of a new cancer therapy using Medical Dictionary for Regulatory Activities (MedDRA)
Time Frame: Up to 2 years
Population: Safety Set Population The Safety Set comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 6
Participants
  Any AE | 6
  Any SAE | 4

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment up to 2 years
Description: AEs and SAEs were collected in Safety Set Population which comprised of all participants who received at least one dose of study treatment.
Arm/Group | Cohort A
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=6)
Nausea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Granulomatous liver disease (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=6)
Anaemia (Blood and lymphatic system disorders) | 4
Mitral valve incompetence (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Ocular hypertension (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 4
Chills (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Candida infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Blood lactate dehydrogenase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Lipase increased (Investigations) | 2
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT01978236/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT01978236/SAP_001.pdf